CLINICAL TRIAL: NCT07207616
Title: Level and Determinants of Advanced Life Support Knowledge Among Nurses in Spain and Effectiveness of an Educational Intervention for Nursing.
Brief Title: Level and Determinants of Advanced Life Support Knowledge Among Nurses
Acronym: CEUJI25
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Colegio oficial de Enfermeros y Enfermeras de Castellón (Unknown); Cardenal Herrera University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UCHCEU-UJI25
Record Dates: First submitted 2025-07-14; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Assess the Knowledge of ALS
Keywords: Advanced life support; Continuing education in nursing; Knowledge; Resuscitation
MeSH Terms: interventions — Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ON LINE (Experimental): Using the Google Sites domain (https://sites.google.com/view/intervencion-sva/inicio), this phase was asynchronous, where participants accessed interactive educational materials and a pre-test on ALS. The online phase was designed to explain theoretical content, and a dedicated webpage was created for this purpose. Each enrolled participant was provided with a link to the site via email. Upon accessing the page, participants were guided on the steps they needed to follow to complete this phase properly.
  Interventions: Other: educational intervention for nursing
- IN PERSON (Experimental): A 15-minute brief review of the theoretical content from the online phase was given at the start of this session. The session was then divided into different workshops where participants practiced various ALS techniques. At the end of the in-person session, participants completed a post-test questionnaire in the classroom. The duration of this phase was four hours.
  Interventions: Other: educational intervention for nursing

INTERVENTIONS:
Other: educational intervention for nursing — A quasi-experimental study was carried out between February and October 2023 in the Valencian Community. This non-randomized intervention followed the TREND guidelines and targeted nurses registered in one of the three official nursing colleges of the region. The educational intervention included an asynchronous online phase hosted on a Google Sites platform, where participants accessed interactive learning materials and completed a pre-test. This was followed by a four-hour in-person session that included a brief theoretical review and hands-on workshops practicing various ALS techniques. A post-intervention test was administered immediately afterward. The intervention led to a noticeable improvement in ALS knowledge, demonstrating its effectiveness.
  Other Names: Formative intervention

SUMMARY:
This study evaluated the knowledge of advanced life support (ALS) among general nurses in Spain and examined the effectiveness of an educational intervention to address identified knowledge gaps. Initially, a cross-sectional study was conducted between November 2020 and February 2021, involving 888 general nurses from all 52 Spanish provinces. Data were collected through a structured self-administered questionnaire assessing demographics, education, professional background, and theoretical ALS knowledge. The results showed that 72.3% of nurses did not achieve the minimum passing score of 70%, revealing significant knowledge deficits, particularly in fluid therapy, defibrillation protocols, ALS algorithms, and use of the LUCAS® CPR device. Higher knowledge levels were associated with female gender, possession of a Master's degree or higher, working in high-risk areas for cardiac arrest, and recent ALS training.

To address these gaps, a second, quasi-experimental study was carried out between February and October 2023 in the Valencian Community. This non-randomized intervention followed the TREND guidelines and targeted nurses registered in one of the three official nursing colleges of the region. The educational intervention included an asynchronous online phase hosted on a Google Sites platform, where participants accessed interactive learning materials and completed a pre-test. This was followed by a four-hour in-person session that included a brief theoretical review and hands-on workshops practicing various ALS techniques. A post-intervention test was administered immediately afterward. The intervention led to a noticeable improvement in ALS knowledge, demonstrating its effectiveness.

Overall, the study highlights insufficient ALS knowledge among Spanish nurses and the need for continuous, structured education. The successful outcome of the intervention reinforces the importance of ongoing training programs to enhance the preparedness of nurses in responding to cardiac arrest and other high-risk clinical scenarios.

DETAILED DESCRIPTION:
Study design, area, and period A cross-sectional study was conducted from November 2020 to February 2021. The study population comprised nurses affiliated with all the official nursing associations in Spain, which are integrated at the national level in the General Council of the Official Nursing Associations of Spain (Consejo General de Colegios Oficiales de Enfermería de España). In this country, membership of one of these official nursing associations is compulsory for the practice of the profession. At the time of the study, the total number of registered nurses in Spain was 291,297.18 The actual sample size for the study was calculated using QuestionPro (https://www.questionpro.com/es/calculadorade-muestra.html#calculadora_de_muestra), considering a target population of 291,297 registered nurses in Spain, a confidence level of 95%, a margin of error of 5%, and an estimated missing rate of 15%. The calculated sample size was 443. A snowball sampling was applied. Data were collected consecutively for each nurse included, as all nurses willing to participate and meeting the study's inclusion criteria participated.

A structured self-administered questionnaire was used for data collection. This questionnaire contained three demographic questions, two questions related to professional experience, five questions regarding educational and ALS training background and professional experience, and 29 theoretical knowledge questions.

The set of 29 theoretical knowledge questions and their respective answer options are derived from a 30-item ERC test (see Supplemental material). This type of test is used in the training courses and assessment of nursing professionals to ensure an adequate level of knowledge of recommended best practice in emergency situations. Given the context, it was determined that a pretest of the instrument would not be conducted. Nevertheless, to avoid information bias, a validation of the content of our adapted and updated Spanish version of the test was conducted by a group of judges (n = 13) with experience in ALS.

For the second phase, a quasi-experimental study was designed between February and October 2023 in the Valencian Community. It was a non-randomized design with an educational intervention and pre-post intervention knowledge evaluation, following the TREND standard guidelines. The study population consisted of nurses registered with one of the three official nursing colleges in the Valencian Community, integrated at the regional level into the Nursing Council of the Valencian Community (CECOVA). At the time of the study, the total number of registered nurses in the Valencian Community was 21,265.

The study reached out to the Nursing Colleges of Castellón, Valencia, and Alicante via email to request their assistance in distributing the questionnaire among their members. Additionally, due to geographic availability, the Colleges of Castellón and Valencia were asked to provide their facilities for the educational intervention. The colleges agreed to distribute the questionnaire, sending the information to their members via email and through their official social media channels. Furthermore, the Castellón and Valencia colleges agreed to provide their facilities and materials for the educational intervention.

Due to challenges in recruiting participants for the in-person phase, contact was made with the Health Sciences Faculties of both the CEU Cardenal Herrera University of Castellón and Jaume I University of Castellón. Both institutions agreed to allow the use of their facilities and to disseminate the study among their employees.

The in-person educational intervention sessions took place at four different locations to facilitate participant attendance.

A non-probabilistic snowball sampling technique was used. The educational intervention was structured into two phases:

Online Phase: Using the Google Sites domain (https://sites.google.com/view/intervencion-sva/inicio), this phase was asynchronous, where participants accessed interactive educational materials and a pre-test on ALS. The online phase was designed to explain theoretical content, and a dedicated webpage was created for this purpose. Each enrolled participant was provided with a link to the site via email. Upon accessing the page, participants were guided on the steps they needed to follow to complete this phase properly.

In-person Phase: A 15-minute brief review of the theoretical content from the online phase was given at the start of this session. The session was then divided into different workshops where participants practiced various ALS techniques. At the end of the in-person session, participants completed a post-test questionnaire in the classroom. The duration of this phase was four hours.

Content of the Intervention:

Online Phase:

Pre-test questionnaire.

Reading theoretical content (CPR).

Solving interactive clinical cases.

Responding to the post-test (for those who did not attend the in-person phase). The estimated duration of this phase was about four hours. The pre- and post-tests were identical and consisted of 19 theoretical knowledge questions. These questions were derived from the 30-item ALS test, available in English (Appendix III). This type of test is used in training courses by the institution to ensure an adequate level of knowledge of best practices in emergency situations. For this study, the test was translated into Spanish and validated by 13 experts (judges) to prevent information bias. The profile of these judges and their recommendations are shown in Table 1. The interactive cases were created using the CANVA application. Furthermore, to ensure the validity of the test, the Cronbach's alpha coefficient for the instrument was determined, yielding a value of 0.670. The survey questionnaires were administered using Microsoft Forms, a survey management software, which was used to create and distribute the questionnaires.

In-person Phase: At the start of this phase, there was a brief 15-minute review of the theoretical content from the online phase. The session was then divided into various workshops where participants practiced different ALS techniques:

Intraosseous Access Workshop: Participants were introduced to the different materials and practiced the intraosseous access technique.

Arrhythmias Workshop: Using a CPR mannequin and a free arrhythmia simulator for PC (Arrhythmia Simulator), participants practiced integrated ALS scenarios.

Airway Management Workshop: Participants practiced endotracheal intubation techniques and familiarized themselves with different supraglottic devices as alternatives for intubation.

Final Scenario: Participants were divided into groups and tasked with integrating all previously learned content into a single clinical case that they had to resolve collectively.

Teaching Methods:

The first phase was conducted online, with the creation of a website using the Google Sites domain. The second phase took place in-person at the Official Nursing Colleges of Castellón and Valencia, as well as at CEU Cardenal Herrera University and Jaume I University.

ELIGIBILITY:
Inclusion Criteria:

* active nursing professionals in the healthcare sector in the Valencian Community, including those working in care, management, teaching, and research roles.
* provide written informed consent before participating in the study.

Exclusion Criteria:

* Nurses who were not registered with an Official Nursing College in the Valencian Community

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
To determine the level of knowledge of nurses in Spain regarding Advanced Life Support (ALS) and identify the factors that influence it. | 6 hours
  the study aims to assess the knowledge of ALS among general nurses in Spain and to identify the socio-educational and occupational factors influencing knowledge.
To assess the effectiveness of an educational intervention aimed at addressing the identified knowledge gaps in ALS. | 4 hours
  the study aims to assess the effectiveness of an educational based in the identified gaps in ALS among general nurses in Spain.

SECONDARY OUTCOMES:
To evaluate knowledge of ALS concepts and techniques. | 30 minutes
  the study aims to evaluate knowledge of ALS concepts based on ERC recommendations.
To identify knowledge gaps in ALS. | 30 minutes
  the study aims to identify knowledge gaps in ALS according to the ERC recommendations.
To determine the sociodemographic, occupational, and educational background characteristics that influence the level of knowledge about ALS. | 30 minutes
  the study aims To determine the sociodemographic, occupational, and educational background characteristics that influence the level of knowledge about ALS based on the ERC recommendations.
To establish the effectiveness of using in-person clinical simulation as a complementary training strategy to online ALS education. | 4 hours
  the study aims to establish the effectiveness of using in-person clinical simulation as a complementary training strategy to online ALS education based on ERC recommentations.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Sanchez-Thevente, phD, Study Director — Cardenal Herrera University
Locations (1):
- Isabel Almodóvar Fernández, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes
There is a first article published at SAGE OPEN MEDICINE: Level and determinants of advanced life support knowledge among nurses in Spain: A national cross-sectional study
Supporting Information: CSR
Time Frame: November 2020 - October 2023
URL: https://journals.sagepub.com/doi/10.1177/20503121251326655